CLINICAL TRIAL: NCT02773680
Title: Assessment of CT-derived Thoracic Electrical-Impedance-Tomography Finite Element Models
Brief Title: Human Electrical-Impedance-Tomography Reconstruction Models
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ass.-Prof. Dr. Stefan Boehme, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1917/2015
Record Dates: First submitted 2016-05-09; First posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Respiratory Monitoring
Keywords: respiration; monitoring, physiologic; diagnostic techniques, respiratory system
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study cohort 1 (Experimental): "electrical impedance tomography"
  Interventions: Device: "electrical impedance tomography"

INTERVENTIONS:
Device: "electrical impedance tomography" — One continous electrical impedance tomography (EIT) measurement per subject of approximately 5 minutes duration (2 min prior to MDCT scanning, during end-inspiratory MDCT acquisition and 2 min after MDCT scanning)

SUMMARY:
Current EIT analyses are based on the assumption of a circular thorax-shape and do not provide any information on lung borders. The aim is to obtain the body and lung border contours of male subjects by multi-detector computed tomography (MDCT) in defined thresholds of anthropometric data (gender = male; height; weight) for calibration of more realistic EIT reconstruction models.

DETAILED DESCRIPTION:
A major drawback of EIT is its relatively poor spatial resolution and its limitation in measuring changes in bioimpedance as compared to a reference state (and not absolute quantities). Therefore, the technique cannot differentiate between extrapulmonary structures (muscles, thorax, heart, large vessels, spine, etc.) and non-aerated lung tissues - which is a major limitation for the clinical use of information derived from EIT-imaging. Moreover, current EIT-reconstruction algorithms are based on the consideration of a complete circular thoracic shape and do not take into account the body contours and lung borders.

The investigators are convinced that EIT-derived dynamic bedside lung imaging can be advanced by morphing computed tomography (CT) scans of the respective thoracic levels with concomitant EIT images - thus enhancing EIT-image information with CT-data. Integrating the anatomy of thoracic shape and lung borders provided by high-spatial resolution multi detector CT-scans (MDCT) with high-temporal resolution EIT has the potential to improve image quality considerably. This data can be used to compute mean EIT-reconstruction models that further offer the possibility to develop novel and clinically meaningful EIT parameters.

Therefore, the investigators hypothesize that by integration of CT-scan information of body and lung contours (and by computing different EIT reconstruction models) the current methodological limitations of EIT technology can be overcome.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous breathing male subjects
* age > 18,
* clinical indication for thoracic CT scanning,
* matching of weight and height to the predefined model-thresholds

Exclusion Criteria:

* pre-existing chronic pulmonary disease
* skin lesions / wounds in the thoracic plane where the EIT SensorBelt will be attached
* known allergy against any ingredient of the used ContactAgent
* abnormalities in thoracic shape as defined by the radiologist in charge (e.g. extreme kyphosis, funnel chest, pigeon breast, multiple rip fractures)
* pneumothorax
* pace maker (external and internal)
* other implanted electrical devices
* other methods measuring bioimpedance

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-11 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Electrical Impedance Tomography Finite Element Model | approximately 1 year through study completion
  Based on CT-derived thorax, lung and heart contours we propose to calculate human finite element models (FEM) for EIT analysis

SECONDARY OUTCOMES:
height | at the time-point of inclusion
weight | at the time-point of inclusion
gender | at the time-point of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Boehme, MD, Principal Investigator — Department of General Anesthesia, Intensive Care Medicine and Pain Management, Medical University of Vienna, Austria

IPD SHARING:
Plan to Share IPD: No